CLINICAL TRIAL: NCT01619150
Title: A Single Center, Randomized, Double-blind, Placebo-controlled 2-way Crossover Study to Investigate the Mechanism of Action of Etoricoxib in Subjects With Osteoarthritis Knee Pain.
Brief Title: A Single Center 2-way Crossover Study to Investigate the Mechanism of Action of Etoricoxib in Subjects With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C4Pain (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OSKNEEPA02
Record Dates: First submitted 2012-06-07; First posted 2012-06-14 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Osteoarthritis
Keywords: knee; osteoarthritis; central sensitization; mechanical detection; pain threshold; quantitative sensory testing; pain biomarkers; COX-2 inhibitors; etoricoxib.
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib, followed by placebo (Other): 4 weeks of treatment with etoricoxib, followed by a wash out period of at least 6 days, followed by another 4 weeks of treatment with placebo.
  Interventions: Drug: Etoricoxib, followed by placebo (matching tablet, without active ingredient)
- Placebo, followed by etoricoxib (Other): 4 weeks of treatment with placebo, followed by a wash out period of at least 6 days, followed by another 4 weeks of treatment with etoricoxib.
  Interventions: Drug: Placebo (matching tablet, without active ingredient), followed by etoricoxib

INTERVENTIONS:
Drug: Etoricoxib, followed by placebo (matching tablet, without active ingredient) — Sequence 1: 1 tablet of 60 mg etoricoxib daily for 4 weeks, for oral use. Sequence 2: 1 tablet of matching placebo daily for 4 weeks, for oral use.
  Other Names: Acoxia®
  Arms: Etoricoxib, followed by placebo
Drug: Placebo (matching tablet, without active ingredient), followed by etoricoxib — Sequence 1: 1 tablet of matching placebo daily for 4 weeks, for oral use. Sequence 2: 1 tablet of 60 mg etoricoxib daily for 4 weeks, for oral use.
  Other Names: Acoxia®
  Arms: Placebo, followed by etoricoxib

SUMMARY:
The purpose of this study is to investigate which pain mechanisms that can be affected by etoricoxib compared to placebo (inactive medication)in subjects with painful knee osteoarthritis af 4 weeks of treatment.

DETAILED DESCRIPTION:
Study Rationale: The purpose of this study is to investigate which pain mechanisms in subjects with painful knee osteoarthritis can be affected by the peripheral and central actions of etoricoxib as compared to placebo during a 4 week treatment therapy period.

The present study will utilize a set of quantitative mechanism based pain biomarkers to assess peripheral and central pain manifestations in OA and the influence of etoricoxib on those individual manifestations in an attempt to understand and explain clinical pain alleviation.

Study Treatment: Subjects will be randomized to one of the 2 sequences of treatment: Sequence 1 (60 mg/day etoricoxib followed by placebo) or Sequence 2 (placebo followed by 60 mg/day etoricoxib). The two treatment periods of 4 weeks each are separated by a washout period of at least 6 days.

Primary Objective: To assess which pain mechanisms are modulated by 60 mg daily administration of etoricoxib compared to placebo in subjects with osteoarthritic (OA) knee pain during two treatment periods of 4-weeks each.

Secondary Objectives: To evaluate if changes in any of the mechanism based experimental pain assessment parameters can explain changes in clinical outcome parameters.

To profile drug responders- versus non-responders based on pain mechanisms involved.

To investigate if change in inflammatory, bone and cartilage related bio-chemical biomarkers can explain changes in either experimental or clinical pain parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IRB/IEC specific) has been obtained prior to initiation of any protocol required procedures.
2. Male or female between 40 and 75 years of age. Females of childbearing potential must have a negative urine pregnancy test at screening.
3. Body weight >40 kg and <150 kg with a body mass index (BMI) between 19-40 kg/m2 inclusive.
4. Idiopathic osteoarthritic knee pain diagnosed in accordance with the American College of Rheumatology modified clinical classification criteria (Altman et al, 1986) and verified radiologically as Kellgren-Lawrence grade I, II or III (Kellgren and Lawrence, 1957) at the index knee. The clinical diagnosis of OA will be confirmed by the ACR clinical and radiographic criteria for classification of idiopathic OA based upon the following criteria (index knee):

   1. Knee pain for at least 14 days per month for the 3 months before study entry.
   2. Osteophytes (with radiographic evidence).
   3. And at least 1 of the following 3 conditions: Age >50, or morning stiffness <30 minutes, or crepitus.
   4. X-ray images of the knee joints are available confirming OA. X-ray images older than12 months cannot be used. New photos are needed to confirm the diagnostic criteria for OA.
5. For the index knee, the average of the worst daily pain score over the last 14 days prior to day 0 must be 4.0 to 9.0. The 14-day average score will be derived from worst daily pain scores recorded in a diary for the index knee.
6. Discontinued use of all analgesic medications (including over-the-counter analgesics/ Non-Steroidal Anti-Inflammatory Drug at least 3 days prior to visit 2 (subjects are allowed limited use of analgesic medications).
7. Have agreed to maintain the same activity level throughout the course of the study.

Exclusion Criteria:

1. Have a history of recurrent seizures other than febrile seizures.
2. Have a history of frequent and/or severe allergic reactions with multiple medications.
3. Have a current or recent history, as determined by the investigator or his delegates, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, psychiatric or cerebral disease which could interfere with the subject's participation in the study.
4. At screening, have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participation in the study. In addition, subjects with following findings will be excluded:

   1. Confirmed Bazett's corrected QT (QTcB) interval > 450 msec for men and > 470 msec for women at screening. If QTcB is prolonged a second ECG will be taken to confirm the finding; (additional ECGs may be performed if required),
   2. Bundle branch blocks and other conduction abnormalities other than mild first degree atrio-ventricular block, left anterior hemi block due to left axis deviation and right bundle branch block of benign origin i.e. not caused by other cardiac disease,
   3. Irregular rhythms other than sinus arrhythmia or occasional supraventricular or ventricular ectopic beats,
   4. History of unexplained syncope,
   5. Family history of unexplained sudden death or sudden death due to long QT syndrome,
   6. T-wave configurations are not of sufficient quality for assessing QT interval determination, as assessed by the investigator.
5. Have an alanine aminotransaminase > 2.5 times Upper Limit of Normal (ULN) at screening, based on reference ranges of the local laboratory. Moderate or greater hepatic impairment.
6. Have prior renal transplant, current renal dialysis or severe renal insufficiency (determined by a derived glomerular filtration rate using Cockcroft Gault formula of ≤30 ml/min/1,73m² calculated by the local lab), or serum creatinine laboratory value >1.5 times ULN, based on the reference ranges of the local laboratory.
7. Have active peptic ulcer or gastrointestinal bleeding.
8. Have known inflammatory intestinal disease.
9. Subject with ischemic heart disease, peripheral arterial disease and/or cerebrovascular disease.
10. Subject with congestive heart failure (NYHA II-IV).
11. Subject with uncontrolled arterial hypertension (>160/90).
12. Subject with diabetes mellitus and documented atherosclerosis.
13. History of bronchospasms, acute rhinitis, nasal polyps, angioneurotic edema, urticaria or other type of allergic reaction after having used acetylic acid or NSAID, inclusive COX-2 inhibitors.
14. Is allergic to the active ingredient of etoricoxib or one or more of the excipients.
15. Pregnant female, breast feeding or planning a pregnancy during the study period. Females of child-bearing potential, not using a reliable means of contraception.
16. Subject with an active malignancy of any type or a history of malignancy within the last 5 years (except basal cell carcinoma of the skin that has been excised prior to study start).
17. Are taking any excluded medications (analgesic medications) that cannot be discontinued during the screening period (3 days prior to visit 2).
18. Subject in treatment with anticoagulants (with the exception of acetylsalicylic acid), methotrexate or rifampicin or antihypertensives (with the exception of Ca+-antagonists).
19. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at Visit 1.
20. Have a history of substance abuse or dependence within the past year, excluding nicotine and caffeine.
21. Subject at a high risk of infection (e.g. leg ulcers, indwelling urinary catheter and persistent or recurrent chest infections and subjects who are permanently bed ridden or wheelchair bound).
22. Subject with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis).
23. Have an autoimmune disorder (not including psoriasis).
24. Subject that do not fully understand the EPM procedures according to investigator experience.
25. Investigator site personnel directly affiliated with this study and/or their immediate family cannot participate. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
26. Subject diagnosed with any condition suggestive of a secondary cause of knee OA including but not limited to knee trauma, septic arthritis, inflammatory joint disease, articular fracture, major dysplasia or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, or primary osteochondromatosis.
27. History of surgery (including arthroscopy) in the index knee within 3 months prior to visit 1 or already planned surgery of the index knee at any time.
28. History of significant prior injury to the index knee within 12 months prior to visit 1.
29. Subject diagnosed with Kellgren and Lawrence grade IV at the index knee.
30. Use of lower extremity assistive devices other than a knee brace or 'shoe lift'. Use of a cane in the hand opposite to the index knee is acceptable.
31. History of prior synovial fluid analysis showing a White Blood Cell count ≥ 2000 mm3 that is indicative of a diagnosis other than OA at the index knee.
32. Have a confounding painful condition that may interfere with assessment of the index knee joint. (Knee pain should be the predominant pain. Mild OA of the hands is allowed, for instance).
33. History of any other musculoskeletal or arthritic condition that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study (i.e., currently symptomatic fractures or any concurrent rheumatic disease such as but not limited to fibromyalgia, rheumatoid arthritis, gout, pseudo-gout or Paget's disease and Reiter's syndrome are excluded).
34. Have used corticosteroids prior to baseline:

    1. Intra-articular injection of steroids into the index knee or into any other site than the index knee within the previous 3 months,
    2. Intra-muscular corticosteroid injections within the previous 3 months,
    3. Oral corticosteroids within the previous 1 month.
35. Have initiated or changed their established physiotherapy program within the last 14 day prior to visit 3.
36. Have not recorded a minimum of 10 days of diary data of the last 14 days immediately preceding visit 3.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in Experimental mechanism based Pain Measures (EPMs)during two treatment periods of 4-weeks each | The EPMs will be measured: at V3, prior to 1. treatment sequence w/ Medication/Placebo; at V5, after 4 weeks of treatment; at V6, prior to 2. treatment sequence w/ Medication/Placebo; at V8, after 4 weeks of treatment.
  The following EPMs will be applied:
  * Quantitative Sensory Testing (QST) of 3 knee joint pain locations
  * Spreading sensitization
  * Pain areas
  * Wind-up like pain
  * Descending noxious inhibitory control
  * Cuff evoked pain
  * Infrared thermography of both knees

SECONDARY OUTCOMES:
Change in Clinical Outcome measures during two treatment periods of 4-weeks each | The Clinical Outcome measures will be measured at screening and throughout the two treatment sequences. The study period is in total 16 weeks. Some measures will be recorded daily, others only at study visits.
  Change of pain severity as measured by the daily 24-hour average pain score (APS), night pain and worst daily pain, the following questionnaires: PQAS, BPI, IGIC, PGAC, WOMAC, Dolotest® and PDQ. Furthermore time and pain intensity from a 40 m self-paced walk test and from a 11 step stair climb test.
  Fasting plasma, serum and urine samples will be collected and stored for potential further analysis of e.g. IL-6, IL-8, CTX1, CTX2, TNFα, CCL2, CO1, CO2, sCRP, CRP25, C1M, C2M, C3M, OC, MMP.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Hoeck, MD PhD, Study Director — C4Pain
Locations (1):
- CCBR A/S, Aalborg, Aalborg, Denmark

REFERENCES:
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Brooks P, Kubler P. Etoricoxib for arthritis and pain management. Ther Clin Risk Manag. 2006 Mar;2(1):45-57. PMID 18360581
- [Background] Cannon CP, Curtis SP, FitzGerald GA, Krum H, Kaur A, Bolognese JA, Reicin AS, Bombardier C, Weinblatt ME, van der Heijde D, Erdmann E, Laine L; MEDAL Steering Committee. Cardiovascular outcomes with etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2006 Nov 18;368(9549):1771-81. doi: 10.1016/S0140-6736(06)69666-9. PMID 17113426
- [Background] Cleeland CS, Nakamura Y, Mendoza TR, Edwards KR, Douglas J, Serlin RC. Dimensions of the impact of cancer pain in a four country sample: new information from multidimensional scaling. Pain. 1996 Oct;67(2-3):267-73. doi: 10.1016/0304-3959(96)03131-4. PMID 8951920
- [Background] Felson DT. Developments in the clinical understanding of osteoarthritis. Arthritis Res Ther. 2009;11(1):203. doi: 10.1186/ar2531. Epub 2009 Jan 30. PMID 19232065
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Freynhagen R, Rolke R, Baron R, Tolle TR, Rutjes AK, Schu S, Treede RD. Pseudoradicular and radicular low-back pain--a disease continuum rather than different entities? Answers from quantitative sensory testing. Pain. 2008 Mar;135(1-2):65-74. doi: 10.1016/j.pain.2007.05.004. Epub 2007 Jun 13. PMID 17570589
- [Background] Graven-Nielsen T, Arendt-Nielsen L. Assessment of mechanisms in localized and widespread musculoskeletal pain. Nat Rev Rheumatol. 2010 Oct;6(10):599-606. doi: 10.1038/nrrheum.2010.107. Epub 2010 Jul 27. PMID 20664523
- [Background] Guy and Bonato (Eds). Manual for the ECDEU Assessment Battery. 2nd revised edition. Chevy Chase, MD: National Institute of Mental Health 1976.
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Jansen JP, Gaugris S, Choy EH, Ostor A, Nash JT, Stam W. Cost effectiveness of etoricoxib versus celecoxib and non-selective NSAIDS in the treatment of ankylosing spondylitis. Pharmacoeconomics. 2010;28(4):323-44. doi: 10.2165/11314690-000000000-00000. PMID 20222755
- [Background] Jespersen A, Dreyer L, Kendall S, Graven-Nielsen T, Arendt-Nielsen L, Bliddal H, Danneskiold-Samsoe B. Computerized cuff pressure algometry: A new method to assess deep-tissue hypersensitivity in fibromyalgia. Pain. 2007 Sep;131(1-2):57-62. doi: 10.1016/j.pain.2006.12.012. Epub 2007 Jan 25. PMID 17257757
- [Background] Kristiansen K, Lyngholm-Kjaerby P, Moe C. Introduction and Validation of DoloTest((R)): a new health-related quality of life tool used in pain patients. Pain Pract. 2010 Sep-Oct;10(5):396-403. doi: 10.1111/j.1533-2500.2010.00366.x. PMID 20384966
- [Background] Lin HY, Cheng TT, Wang JH, Lee CS, Chen MH, Lei V, Lac C, Gammaitoni AR, Smugar SS, Chen WJ. Etoricoxib improves pain, function and quality of life: results of a real-world effectiveness trial. Int J Rheum Dis. 2010 May;13(2):144-50. doi: 10.1111/j.1756-185X.2010.01468.x. PMID 20536599
- [Background] Moore RA, Moore OA, Derry S, McQuay HJ. Numbers needed to treat calculated from responder rates give a better indication of efficacy in osteoarthritis trials than mean pain scores. Arthritis Res Ther. 2008;10(2):R39. doi: 10.1186/ar2394. Epub 2008 Apr 2. PMID 18384679
- [Background] Renner B, Zacher J, Buvanendran A, Walter G, Strauss J, Brune K. Absorption and distribution of etoricoxib in plasma, CSF, and wound tissue in patients following hip surgery--a pilot study. Naunyn Schmiedebergs Arch Pharmacol. 2010 Feb;381(2):127-36. doi: 10.1007/s00210-009-0482-0. Epub 2010 Jan 6. PMID 20052461
- [Background] Staahl C, Christrup LL, Andersen SD, Arendt-Nielsen L, Drewes AM. A comparative study of oxycodone and morphine in a multi-modal, tissue-differentiated experimental pain model. Pain. 2006 Jul;123(1-2):28-36. doi: 10.1016/j.pain.2006.02.006. Epub 2006 Apr 4. PMID 16600508
- [Background] Staahl C, Reddy H, Andersen SD, Arendt-Nielsen L, Drewes AM. Multi-modal and tissue-differentiated experimental pain assessment: reproducibility of a new concept for assessment of analgesics. Basic Clin Pharmacol Toxicol. 2006 Feb;98(2):201-11. doi: 10.1111/j.1742-7843.2006.pto_211.x. PMID 16445596
- [Background] Trelle S, Reichenbach S, Wandel S, Hildebrand P, Tschannen B, Villiger PM, Egger M, Juni P. Cardiovascular safety of non-steroidal anti-inflammatory drugs: network meta-analysis. BMJ. 2011 Jan 11;342:c7086. doi: 10.1136/bmj.c7086. PMID 21224324
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Background] van Spil WE, DeGroot J, Lems WF, Oostveen JC, Lafeber FP. Serum and urinary biochemical markers for knee and hip-osteoarthritis: a systematic review applying the consensus BIPED criteria. Osteoarthritis Cartilage. 2010 May;18(5):605-12. doi: 10.1016/j.joca.2010.01.012. Epub 2010 Feb 6. PMID 20175979
- [Background] You HJ, Morch CD, Chen J, Arendt-Nielsen L. Differential antinociceptive effects induced by a selective cyclooxygenase-2 inhibitor (SC-236) on dorsal horn neurons and spinal withdrawal reflexes in anesthetized spinal rats. Neuroscience. 2003;121(2):459-72. doi: 10.1016/s0306-4522(03)00296-3. PMID 14522004
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771